CLINICAL TRIAL: NCT05529550
Title: Assessment of Nutritional Status and Role of Insulin-like Growth Factor-1 in Children With Thalassemia Major
Brief Title: Assessment of Nutritional Status and Role of Insulin-like Growth Factor-1 in Children
Status: Completed | Type: Observational
Sponsor: Menoufia University (Other)
Responsible Party: Principal Investigator, Samar Abdelhameed, Dr, Menoufia University
Other Study IDs: insulin-like growth factor-1
Record Dates: First submitted 2022-09-02; First posted 2022-09-07 (Actual); Last update posted 2022-09-07 (Actual); Status verified 2022-09

CONDITIONS: Thalassemia
Keywords: Insulin-like growth factor 1
MeSH Terms: conditions — Thalassemia

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients: 67 children in the age group of 2-18 years with confirmed diagnosis of Beta thalassemia major.
- Healthy control: 35 healthy children

SUMMARY:
Many studies done on children with thalassemia have shown a variable prevalence of defective IGF-I concentrations have been shown to be low in the majority of children, with or without GH deficiency. The Aim of this study to assess nutritional status and role of Insulin-like growth factor 1 (IGF-1) and its associating factors in children with thalassemia major

ELIGIBILITY:
Inclusion Criteria:

* Children in the age group of 2-18 years with confirmed diagnosis of Beta thalassemia major.

Exclusion Criteria:

* Children with other chronic diseases (cardiac, renal, vascular)
* Children with malignancy

Ages: 1 Year to 18 Years | Sex: All
Age Groups: Child, Adult
Study Population: 67 Children in the age group of 2-18 years with confirmed diagnosis of Beta thalassemia, and 35 healthy control
Sampling Method: Non-Probability Sample
Enrollment: 102 (Actual)
Dates: Start 2020-10-01 (Actual); Primary Completion 2021-11-01 (Actual); Study Completion 2021-12-01 (Actual)

PRIMARY OUTCOMES:
IGF-1 | at the time of recruitment
  insulin-like growth factor-1 which measured by enzyme linked immunosorbent assay (ELISA).

CONTACTS AND LOCATIONS:
Locations (1):
- Samar Abd El-Hameed, Shibīn al Kawm, Egypt